CLINICAL TRIAL: NCT06808542
Title: Pelvic Floor Dysfunction Among Female Physiotherapy Students: A Cross-Sectional Study
Status: Recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Doaa A. Osman, Principal Investigator, Cairo University
Other Study IDs: P.T.REC/012/005385
Record Dates: First submitted 2025-01-30; First posted 2025-02-05 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Pelvic Floor Disorders
MeSH Terms: conditions — Pelvic Floor Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This study aims to:

1. estimate the prevalence of pelvic floor dysfunction among female physiotherapy students at Cairo University.
2. identify potential risk factors that may be associated with pelvic floor dysfunction in this student population.
3. assess the level of awareness regarding pelvic floor health among female physiotherapy students at Cairo University.
4. explore how female physiotherapy students at Cairo University utilize available healthcare resources for managing pelvic floor-related concerns.

DETAILED DESCRIPTION:
Pelvic floor dysfunction (PFD) is a global health problem that affects millions of women worldwide. It encompasses a broad range of interrelated disorders affecting the pelvic region, including urinary incontinence, pelvic pain, constipation, sexual dysfunction, and pelvic organ prolapse. While PFD is often associated with pregnancy, childbirth, and aging, recent studies suggest that these conditions may also affect younger populations, including nulliparous women.

Pelvic floor health is crucial for supporting pelvic organs, maintaining continence, and facilitating sexual function. However, the impact of PFD on women's health and quality of life is significant, with important consequences for physical and mental well-being. These disorders often coexist and compound each other's impact, leading to disabling symptoms, embarrassment, social isolation, impaired task performance, loss of personal and intimate relationships, and reduced participation in leisure activities.

Despite the substantial burden of PFD, there is a lack of comprehensive data on the prevalence, risk factors, and awareness levels of these conditions among specific populations, particularly young women pursuing higher education. Physiotherapy students, who are expected to have a good understanding of musculoskeletal and pelvic health, represent an important group to study in this context.

ELIGIBILITY:
Inclusion Criteria:

* Virgin undergraduate physiotherapy students.
* Their age will range from 18-25 years.

Exclusion Criteria:

* Neurological disorders or injuries that may affect pelvic floor function (e.g., fibromyalgia and multiple sclerosis).
* Mental health or cognitive disorders that could affect data collection.
* Females who have undergone any form of abdominal surgery prior to the time of the study.
* Females with current use of medications that may affect pelvic floor function (e.g., anticholinergics, opioids, antidepressants).

Ages: 18 Years to 25 Years | Sex: Female
Age Groups: Adult
Study Population: This study aims to enrol a sample of 180 female physiotherapy students from Cairo University, from the first-year to the fifth-year levels, to ensure adequate representation across different stages of the academic program.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2025-02-04 (Actual); Primary Completion 2025-04-04 (Estimated); Study Completion 2025-04-25 (Estimated)

PRIMARY OUTCOMES:
Modified Australian pelvic floor questionnaire | 2 months
  It will be used to estimate the prevalence of pelvic floor disorders through assessing their bladder function, bowel function, and pelvic organ prolapse. This questionnaire will be administered electronically via online survey platforms.

SECONDARY OUTCOMES:
A self-administered survey | 2 months
  A self-administered survey will be used to assess potential associated risk factors, including lifestyle habits, weight, BMI, family history, mental health factors (stress, anxiety, depression), physical health factors (sleep, exercise, dietary habits). Also, it will assess students' awareness of pelvic floor health and their utilization of available healthcare resources for managing pelvic floor-related concerns.

CONTACTS AND LOCATIONS:
Overall Officials: Doaa A. Osman, PhD, Study Chair — Assistant Professor, Cairo university
Locations (1):
- Cairo University, Giza, Egypt